CLINICAL TRIAL: NCT05078450
Title: Mood Lifters Online
Brief Title: Mood Lifters Online for Graduate Students and Young Professionals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Patricia Deldin, Professor of Psychology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00163570
Record Dates: First submitted 2021-09-22; First posted 2021-10-14 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Depression; Anxiety Disorders; Mood Disorders; Mental Illness; Stress
MeSH Terms: conditions — Depression; Anxiety Disorders; Mood Disorders; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Graduate Student Program (Experimental): This is the graduate student version of the program. The original program has been tailored to this population to meet its specific needs and address its specific concerns.
  Interventions: Behavioral: Mood Lifters
- Young Professional Program (Experimental): This is the young professional version of the program. The original program has been tailored to this population to meet its specific needs and address its specific concerns.
  Interventions: Behavioral: Mood Lifters
- Waitlist (No Intervention): This is the waitlist. Participants may be randomly assigned here first. After the typical period fo the intervention on the waitlist (12 weeks), these participants will be invited to join the arm which they are most appropriate for (i.e., graduate student or young professional).

INTERVENTIONS:
Behavioral: Mood Lifters — Participants will need to attend 12 hour long virtual weekly meetings on Zoom that focus on helpful mental health strategies and skills. Participants will be encourage to practice what they learn at home in order to improve their mood or mental wellness.
  Arms: Graduate Student Program; Young Professional Program

SUMMARY:
Mood Lifters is a revolutionary mental wellness program that teaches scientifically validated strategies in a supportive group setting. This study will test two new versions of the program designed specifically for graduate students and young professionals.

Participants will need to attend 12 hour long virtual weekly meetings on Zoom that focus on helpful mental health strategies and skills. Participants will be encourage to practice what the participants learn at home in order to improve their mood or mental wellness. Additionally, participants will complete a series of measures (approx. 1-1.5 hours) prior to, at the end of the program, 1 month after the program and 6 months after the program.

ELIGIBILITY:
Inclusion Criteria:

* Participants ages 22-32 (must identify as either a graduate student or a young professional)

Exclusion Criteria:

* Active suicidality, mania, or psychosis

Ages: 22 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 362 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire - 9 | through study completion, an average of 1 year
  Assesses Depressive Symptoms (Range 0-27; higher scores indicate more significant symptoms of depression)
Generalized Anxiety Disorder - 7 | through study completion, an average of 1 year
  Assesses Anxiety Symptoms (Range 0-21; higher scores indicate more significant symptoms of anxiety)
Perceived Stress Scale | through study completion, an average of 1 year
  Assesses Perceived stress (Range 0-40; higher scores indicate more significant perceived stress)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garg T, Votta CM, Prakash N, Deldin PJ. An investigation into the effectiveness of Mood Lifters in the context of trauma exposure. Psychol Serv. 2024 Aug;21(3):518-528. doi: 10.1037/ser0000789. Epub 2023 Aug 24. PMID 37616078
- [Background] Pokowitz EL, Prakash N, Planaj D, Oprandi S, Deldin PJ. Mood Lifters for Graduate Students and Young Adults: A Mixed-Methods Investigation into Mechanisms of Change in Online Group Therapy. Behav Sci (Basel). 2024 Mar 20;14(3):252. doi: 10.3390/bs14030252. PMID 38540555
- [Background] Prakash N, Votta CM, Deldin PJ. Treatment for graduate students: Blunting the emotional toll of postgraduate education. J Consult Clin Psychol. 2023 Dec;91(12):708-716. doi: 10.1037/ccp0000844. Epub 2023 Sep 21. PMID 37732972